CLINICAL TRIAL: NCT01108003
Title: Pilot Pre-cystectomy Trial of Broccoli Extract in Patients With Superficial or Locally Advanced Bladder Cancer
Brief Title: Broccoli Sprout Extract in Treating Patients With Transitional Cell Bladder Cancer Undergoing Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low accrual
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Johns Hopkins University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 129408; NCI-2010-00759
Record Dates: First submitted 2010-04-19; First posted 2010-04-21 (Estimated); Results first posted 2016-06-23 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-05

CONDITIONS: Recurrent Bladder Cancer; Stage 0 Bladder Cancer; Stage I Bladder Cancer; Stage II Bladder Cancer; Transitional Cell Carcinoma of the Bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive oral broccoli sprout extract once daily on days 1-14 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: broccoli sprout extract; Other: laboratory biomarker analysis
- Arm 2 (Placebo Comparator): Patients receive mango juice alone.
  Interventions: Other: Mango Juice

INTERVENTIONS:
Drug: broccoli sprout extract — Given orally
  Arms: Arm I
Other: laboratory biomarker analysis — Correlative studies
  Arms: Arm I
Other: Mango Juice — given orally
  Arms: Arm 2

SUMMARY:
Rationale: Broccoli sprout extract contains ingredients that may prevent or slow the growth of certain cancers.

Purpose: This pilot study is studying the side effects of broccoli sprout extract in treating patients with transitional cell bladder cancer undergoing surgery.

DETAILED DESCRIPTION:
Primary Objectives:

I. To determine the tolerability and toxicity of a broccoli sprout extract (providing 200 micro mol isothiocyanate/dose/per day) given for 14 days in patients destined to undergo definitive bladder resection for bladder cancer.

Secondary Objectives:

I. Establish the safety of administration of the broccoli extract on the bladder surgery specifically.

II. Determine the levels of isothiocyanates and their metabolites in urine, blood, benign urothelium and bladder cancer tissue.

III. Assess the antitumor effects of broccoli extract on the primary bladder tumor by measuring angiogenesis, cell proliferation and apoptosis.

IV. Determine the feasibility of treating patients with 200 micro mol isothiocyanate per dose per day of broccoli sprout extract in future therapeutic and prevention clinical trials.

Outline: Patients receive oral broccoli sprout extract once daily on days 1-14 in the absence of disease progression or unacceptable toxicity. After completion of study treatment, patients are followed at 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Any patient eligible for superficial bladder cancer
* Patients must be considered fit for surgical resection with curative intent
* No chemotherapy, surgery (excluding transurethral resection of bladder tumor [TURBT], BCG or radiotherapy in the prior 4 weeks [6 weeks for mitomycin C or interferon])
* No previous treatment/ingestion with broccoli extracts
* Eastern Oncology Group (ECOG) performance status 0-2
* AST and ALT =< 2.5 times ULN (upper limit of normal)
* Total bilirubin =< 2.0 mg/dL
* Creatinine Clearance >= 30 ml/min
* WBC > 3000 mm^3
* Absolute neutrophil count > 1000/mm^3
* Platelets > 100,000/mm^3
* All patients must sign a study-specific consent form indicating that they are aware of the investigational nature of this study

Exclusion Criteria:

* Have participated in any clinical trial involving conventional or investigational drugs or devices within the previous 4 weeks
* Prior radiation to the pelvis
* Intractable urinary tract infection that has not responded to antibiotic treatment
* Active, uncontrolled bacterial, viral, or fungal infection including HIV
* Have had major surgery within 4 weeks of starting therapy (not including placement of vascular access device or TURBT)
* Poor medical risk in the opinion of the treating oncologist due to non-malignant systemic disease
* Pregnant or lactating patients: patients must be postmenopausal or practicing an accepted form of birth control; for patients where pregnancy is a possibility, a pregnancy test will be required prior to initiation of therapy
* Have a history of myocardial infarction or angina pectoris/angina equivalent in the last 6 months (the patient may be on anti-anginal medications if the symptoms have been entirely controlled for greater than 6 months), or have uncontrolled congestive heart failure
* Have a history of bleeding disorders or thrombosis; patients on therapeutic doses of anticoagulation (including coumadin or heparins) are not permitted on trial (this exclusion criterion does not include those patients receiving low dose or prophylactic dose anticoagulation [i.e. coumadin 1 mg daily in patients with central intravenous lines])
* Radiotherapy during the course of the trial
* Inability to tolerate proposed treatment or procedures
* Have additional uncontrolled serious medical conditions or psychiatric illness
* Patients with a history of hepatitis (including but not exclusive to viral hepatitis auto-immune or alcoholic)
* Patients with active thyroid disease (patients with hypothyroidism, adequately replaced on a stable dose of thyroid replacement will be allowed on trial)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-04; Primary Completion 2014-09 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Marshall, PhD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I | Arm 2
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm 2 | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 74 (5.3) | 73 (4.9) | 74 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Toxicity as Assessed by National Cancer Institute (NCI) Common Toxicity Criteria Version 3.0
Description: Number of participants with an adverse event.
Time Frame: 14 days
Population: All treated and eligible patients.
Measure: Number; unit: participants
Arm/Group | Arm I | Arm 2
Number analyzed (Participants) | 4 | 3
participants | 4 | 3

2. Secondary Outcome: Apoptosis, Cell Proliferation, and Microvessel Density
Time Frame: 1 year
Population: Due to the study's early termination and low accrual, data were not collected for this assessment.
Arm/Group | Arm I | Arm 2
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm I | Arm 2
Serious Adverse Events (participants affected / at risk) | 2/4 | 1/3
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=4) | Arm 2 (N=3)
Fungaemia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=4) | Arm 2 (N=3)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood albumin decreased (Investigations) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood calcium decreased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (2) | 1 (1)
Blood magnesium increased (Investigations) | 0 (0) | 1 (1)
Cardiac enzymes increased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram abnormal (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (2) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (8) | 3 (3)
Platelet count decreased (Investigations) | 1 (2) | 0 (0)
White blood cell analysis increased (Investigations) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Penile discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to the study's early termination and low accrual, data were not collected for all study objectives assessment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes